CLINICAL TRIAL: NCT06963671
Title: What is the Effect of Low-load Blood Flow Restriction Training in the Nonoperative Rehabilitation of Ulnar-sided Wrist Pain?
Brief Title: Blood Flow Restriction for Ulnar Sided Wrist Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 80801
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ulnar Wrist Pain
Keywords: blood flow restriction
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm will receive the standard of care treatment for ulnar sided wrist pain
- Blood Flow Restriction (Experimental): The Blood Flow Restriction group will receive BFR treatment
  Interventions: Behavioral: Blood Flow Restriction

INTERVENTIONS:
Behavioral: Blood Flow Restriction — The treatment group will receive standard rehabilitation as a home program plus low-load resistance training with BFR application while at the hand therapy clinic for their appointments
  Arms: Blood Flow Restriction

SUMMARY:
The purpose of this study is to determine the strength, pain and functional benefits of early, low-load resistance training with blood flow restriction (BFR) in ulnar-sided wrist pain treated nonoperatively with immobilization for 4-6 weeks. Hypothesis: patients in the BFR group with have improved grip strength and patient reported outcome measure scores compared to the control group.

DETAILED DESCRIPTION:
Patients presenting to the hand therapy or hand surgery clinic who meet inclusion criteria will be screened, consented, and enrolled. This will include administration of the blood flow restriction screening questionnaire.

Patients with non operatively managed ulnar-sided wrist pain, who have been immobilized for at least 4 weeks 0 days, but no more than 6 weeks 6 days, and are referred to Stanford's Hand Therapy clinic, will receive either standard care or a standard care home program with low-load strengthening under a blood flow restricted (BFR) condition during their therapy sessions. Patients will be assigned to groups in simultaneous enrollment in two arms. The control group will receive standard rehabilitation during therapy visits plus a home program that will be dictated based on the associated phase of rehabilitation. The treatment group will receive standard rehabilitation as a home program plus low-load resistance training with BFR application while at the hand therapy clinic for their appointments, both of which will be dictated based on the associated phase of rehabilitation. Therapists will use the OMNI-Resistance Exercise Scale for Rate of Perceived Exertion Active Muscles (OMNI-RES RPE-AM) to grade all strengthening exercises for each individual in both groups. The target RPE-AM for each exercise will be 7-9 by the last set for resistance exercises in both control and treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients (>18 years) undergoing outpatient rehabilitation at Stanford Hand Therapy
* English fluency and literacy
* Able to take informed consent
* Have acute or chronic ulnar-sided wrist pain referred for a course of hand therapy by a physician or advanced practice provider (APP) and were treated with continuous immobilization for 4-6 weeks.
* Score of 3 or less on blood flow restriction screening questionnaire

Exclusion Criteria:

* Concomitant injuries such as upper extremity fractures or other ligamentous injuries
* TFCC surgery in the affected wrist
* Non-compliance with immobilization
* Patients who complete hand therapy at an outside facility
* Score of 4 or more on blood flow restriction screening questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | From enrollment to 6 weeks after initiation of BRF
  Grip Strength as measured by a dynamometer in pounds.

SECONDARY OUTCOMES:
Patient Reported Wrist Evaluation (PRWE) | From enrollment to 6 weeks after initiation of BRF
  The PRWE is a patient-reported outcome measure created to measure wrist pain and disability in activities of daily living. This scale is scored from 0-100, and lower scores indicate better function while higher scores indicate worse function.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No